CLINICAL TRIAL: NCT04443855
Title: Measuring the Effect of WASH Benefits Interventions on Child Development Outcomes at School Age: Follow up of an Efficacy Trial in Rural Bangladesh
Brief Title: WASH Benefits Child Development Follow up
Acronym: WASH-BFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Stanford University (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-19025
Record Dates: First submitted 2020-04-30; First posted 2020-06-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Child Development; Maternal Depression
Keywords: Child Development; WASH; Nutrition
MeSH Terms: interventions — Water Quality; Sanitation; Hand Disinfection; Nutritional Status

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The outcome assessment team is separate from the implementation team, however due to the nature of the interventions there may be intervention contents visible during the assessment. Data analysis will be masked to randomization status of clusters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Water quality (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Water quality
- Sanitation (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Sanitation
- Hand washing (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Hand washing
- Combined WASH (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Water quality, Sanitation, Hand washing (Combined WASH)
- Nutrition (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Nutrition
- Nutrition+ Combined WASH (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Nutrition, Water quality, Sanitation, Hand washing
- Non-intervention (No Intervention): 180 clusters, approx. 1,440 newborns

INTERVENTIONS:
Behavioral: Water quality — Hardware: Free supplies chlorine tablets (Aquatabs; NaDCC) and a safe storage vessel to treat and store drinking water.
  Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the treatment of all drinking water for children < 36 months of age.
  Arms: Water quality
Behavioral: Sanitation — Hardware: Free child potties, sani-scoop hoes to remove feces from household environments, latrine upgrades to a dual pit latrine Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the use of latrines for defecation and the removal of human and animal feces from the compound.
  Arms: Sanitation
Behavioral: Hand washing — Hardware: Hand washing stations, soapy water bottles located at hand washing locations, detergent soap to supply soapy water bottles.
  Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on hand washing with soap at critical times around food preparation, defecation, and contact with feces.
  Arms: Hand washing
Behavioral: Water quality, Sanitation, Hand washing (Combined WASH) — Hardware: Free supplies Aquatabs; (NaDCC) and a safe storage vessel to treat and store drinking water. Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the treatment of drinking water for children < 36 months.
  Hardware: Free child potties, sani-scoop hoes to remove feces from household environments, latrine upgrades to a dual pit latrine. Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the use of latrines for defecation and the removal of human and animal feces from the compound.
  Hardware: Hand washing stations, soapy water bottles, detergent soap to supply soapy water bottles. Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on hand washing with soap at critical times as food preparation, defecation, and contact with feces.
  Arms: Combined WASH
Behavioral: Nutrition — Supplement: Lipid-based Nutrient Supplement (LNS) delivered daily from ages 6 to 24 months.
  Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages modeled on those recommended in the Guiding Principles for Complementary Feeding of the Breastfed Child and the recent UNICEF Program Guide for Infant and Young Child Feeding Practices.General messages will include (1) practice exclusive breastfeeding from birth to 6 months of age and introduce complementary foods at 6 months of age while continuing to breastfeed; (2) continue breast feeding as you did before receiving LNS; (3) provide your child micronutrient-rich foods such as meat, fish, eggs, and vitamin A rich fruits and vegetables; and (4) feed your child at least 2-3 times per day when 6-8 months old and 3-4 times per day when 9-24 months old.
  Arms: Nutrition
Behavioral: Nutrition, Water quality, Sanitation, Hand washing — Each of the interventions described above for Water Quality, Sanitation & Hand washing (Combined WASH) Plus the intervention described above for nutrition.
  Arms: Nutrition+ Combined WASH

SUMMARY:
The purpose of this study is to determine if the effects of individual and combined water, sanitation, hygiene, and nutrition interventions in early childhood on child development and maternal mental health persist into middle childhood. This study is a follow-up assessment of the children and mothers enrolled in the WASH-Benefits Bangladesh study.

DETAILED DESCRIPTION:
Globally, millions of children experience delays in physical health and cognitive development, due to their exposures to poverty and related issues. In low-and middle-income countries, children experience a dis-proportionally high burden of exposure to poverty and related risk factors for delayed development including of poor health and nutrition, inadequate responsive care giving, and a lack of opportunities for early learning. Water, sanitation and hygiene (WASH) interventions have the potential to positively affect the developmental trajectories of children by reducing enteric pathogen infection, improving child health, and altering parental care practices. A recent cluster-randomized controlled trial (cRCT) in Bangladesh (WASH-Benefits, or WASH-B, Clinical Trials.gov Identifier: NCT01590095), found that improvements in WASH or nutrition supported by intensive interpersonal communication, when delivered either individually or in combination, contributed to improvements in child development outcomes at 1 and 2 years of age, and mothers in all intervention groups reported lower depressive symptoms than mothers in the control households.

This follow-up study, funded by the Bill & Melinda Gates foundation, includes assessments of the children and caregivers originally enrolled in the WASH Benefits intervention 5 years following intervention completion, when the children are 5-8 year of age. The original WASH Benefits intervention enrolled pregnant women between May 31, 2012, and July 7, 2013. The goal of this follow-up study is to examine whether the improvements in child development and maternal mental health are sustained when the children are in middle childhood. Our guiding hypothesis is that interventions that showed early impact will continue to improve child and maternal outcomes at this follow-up time period. Investigators will attempt to collect follow-up data from every household originally randomized to one of the 7 arms in the WASH Benefits trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the wash-benefits Bangladesh intervention

Exclusion Criteria:

* No Exclusion criteria

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4932 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Weschler Primary and Preschool Scales of Development 4th edition (WPPSI-IV) | 5 years after intervention completion
  The WPPSI-IV assessment measures cognitive development and general intellectual abilities in children 2 years 6 months to 7 years 7 months of age (2:6-7:7), and includes assessments of both performance and verbal skills.
Executive Functioning | 5 years after intervention completion
  This executive functioning assessment consists of three sub-scales to assess executive functioning in children including verbal memory, visual and non-verbal memory, and memory capacity.
Child Socioemotional Development | 5 years after intervention completion
  Maternal-report questionnaire designed to measure psychological adjustment in children and aims to detect any emotional or behavioural problems.
Fine Motor Development | 5 years after intervention completion
  Manual Dexterity component of Movement Assessment Battery for Children-2 (MABC-2) is a direct assessment tool used to measure fine motor skills in children 3 to 17 years of age.
Academic achievement | 5 years after intervention completion
  The Wide Range Assessment Test (WRAT) assessment is a written and verbal assessment of reading, writing, and math achievement.

SECONDARY OUTCOMES:
Maternal Mental Health | 5 years after intervention completion
  Center for Epidemiologic Studies Depression Scale (20 questions). This scale contains 20 questions asking about the number of days in the past week the respondent has experienced each of the symptoms.
Home environment | 5 years after intervention completion
  The middle childhood HOME includes caregiver report and observational items to assess the quality and quantity of stimulation and support available to the child at home.
School attendance | 5 years after intervention completion
  Parental report
Height-for-Age Z-scores | 5 years after intervention completion
  Child's standing height, standardized to Z-scores using the WHO 2006 growth standards
Weight-for-Height Z-scores | 5 years after intervention completion
  Child's weight and height, standardized to Weight-for-Height Z-scores using the WHO 2006 growth standards

CONTACTS AND LOCATIONS:
Overall Officials: Mahbubur Rahman, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
We will follow as per icddr,b data sharing policy

REFERENCES:
- [Derived] Tofail F, Pitchik HO, Islam M, Khan R, Shoab AK, Akter F, Aktar S, Huda TMN, Rahman M, Winch PJ, Luby SP, Fernald LCH. Effects of early water, sanitation, handwashing, and nutrition interventions on child development at school age: a follow-on study of a cluster-randomized trial in rural Bangladesh. PLoS Med. 2025 Dec 16;22(12):e1004793. doi: 10.1371/journal.pmed.1004793. eCollection 2025 Dec. PMID 41401135